CLINICAL TRIAL: NCT03523234
Title: Neoadjuvant Therapy Combined With Radical Surgery for the Treatment of Small Cell Lung Cancer (SCLC) in II and IIIA Stage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peng Zhang (Other)
Responsible Party: Sponsor-Investigator, Peng Zhang, director of science and education department, Shanghai Pulmonary Hospital, Shanghai, China
Organization: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: k18-066
Record Dates: First submitted 2018-04-11; First posted 2018-05-14 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Small-cell Lung Cancer
Keywords: neoadjuvant therapy; surgery
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Neoadjuvant Therapy; Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- surgery group (Experimental)
  Interventions: Drug: neoadjuvant chemotherapy; Procedure: radical surgery for stage II and IIIA small cell lung cancer (SCLC); Procedure: prophylactic cranial irradiation; Drug: Chemotherapy
- control group (Placebo Comparator)
  Interventions: Procedure: prophylactic cranial irradiation; Drug: Chemotherapy

INTERVENTIONS:
Drug: neoadjuvant chemotherapy — etoposide with cisplatin/carboplatin, undergoing in prior to the surgery
  Arms: surgery group
Procedure: radical surgery for stage II and IIIA small cell lung cancer (SCLC) — Lobectomy/total lung resection plus mediastinal lymph node dissection.
  Arms: surgery group
Procedure: prophylactic cranial irradiation — prophylactic cranial irradiation (PCI) undergoing with adjuvant chemotherapy simultaneously
Drug: Chemotherapy — etoposide with cisplatin/carboplatin

SUMMARY:
The main purpose of this study is to compare the effects of neoadjuvant with radical surgery on the prognosis of patients with stage II and IIIA small cell lung cancer (SCLC). The primary endpoint of this study is to observe 5-year survival, disease-free survival (DFS), and overall survival (OS) in patients. Secondary efficacy indicators include recurrence rate, surgical complications, resection rate, quality of life (QoL), and exploration biomarker (tumor tissue).

This is a two-arm, open, multicentral clinical study designed to assess the disease-free survival (DFS) and overall survival (OS) of neoadjuvant chemotherapy plus radical surgery for stage II and IIIA small cell lung cancer (SCLC). About 300 patients will be enrolled in the study and randomly divided into two groups of 150 individuals. The neoadjuvant with radical surgery group received 2 to 4 cycles of neoadjuvant treatment with etoposide plus cisplatin/carboplatin before receiving radical surgery, followed by 2 to 4 cycles of adjuvant chemotherapy (etoposide with cisplatin/carboplatin) plus radiotherapy. Patients in the control group are planned to receive 4 to 6 courses of etoposide plus cisplatin/carboplatin for chemotherapy and radiotherapy.

DETAILED DESCRIPTION:
Before chemotherapy is widely used in clinical work, surgery is the main method for the treatment of lung cancer. However, the prognosis of patients with small cell lung cancer (SCLC) is significantly worse than that of other histological types of lung cancer. The only two prospective studies comparing the surgery with other treatments (surgery vs. radiotherapy alone; induction chemotherapy + surgery vs. chemotherapy + radiotherapy) found that patients in surgery group had a poorer prognosis. Thus, small cell lung cancer was determined to be a non-surgically treated disease. Therefore, for patients with stage II and III A SCLC, combined radiotherapy and chemotherapy are currently recommended. The first-line chemotherapy regimens are etoposide plus cisplatin and carboplatin. Surgical treatment is currently only recommended for very early stage SCLC (T1-2N0M0) with postoperative adjuvant chemotherapy, but these patients only account for about 5% of all SCLC patients. Despite the sensitivity to chemotherapy, the long-term survival of small cell lung cancer remains unsatisfactory. For patients with limited SCLC, even if combined with local radiotherapy, there are still 1/4 to 1/3 of patients progressing due to recurrence of local lesions. So the status of surgical treatment is expected to be reassessed. In recent years, retrospective analysis results of some large databases in Europe and the United States have provided a basis for the role of surgery in the treatment of small cell lung cancer (SCLC). It is believed that surgery should be used as one of the treatment options for SCLC. Based on the results of prospective studies and retrospective studies, a well-designed, phased, prospective study is urgently needed to explore the role of surgery in the treatment of SCLC.

In neoadjuvant therapy combined with radical surgery, neoadjuvant chemotherapy is based on the combination of etoposide and cisplatin/carboplatin. Doses of the drugs are taken from the NCCN guideline for the recommended adjuvant chemotherapy for the limited-period SCLC: namely etoposide 120 mg/m2 through intravenous infusion on Day 1, 2, and 3; cisplatin 60 mg/m2 through intravenous infusion on Day 1 (or carboplatin where area under the curve AUC = 5-6); 4 weeks for a cycle, with a total of 2 cycles of neoadjuvant chemotherapy. Radical surgery is performed according to the growth of SCLC patients after neoadjuvant chemotherapy, using lobectomy or pneumonectomy combined with mediastinal lymph node dissection or sampling. 4 weeks after surgery, chemotherapy and concurrent radiotherapy will be performed. The chemotherapy regimen is the same with that of neoadjuvant chemotherapy, with 4 weeks as a cycle and a total of 2 to 4 cycles. Radiotherapy and adjuvant chemotherapy are planned to be started synchronously, the patients whose intraoperative pathology showed no lymph node metastasis (N0) will receive prophylactic brain irradiation (PCI) treatment and adjuvant chemotherapy synchronously. Within 10 days, the patients will receive a total dose of 25 Gy of PCI, once a day, 2.5 Gy of brain irradiation each time. The patients whose intraoperative pathology show that there is lymph node metastasis (N1-2) are planned to receive PCI combined with mediastinal radiation therapy: namely the patient receive a total of 45 Gy within 3 weeks at the start of adjuvant chemotherapy, twice a day, 1.5 Gy of chest irradiation each time, and the PCI treatment is the same with patients whose intraoperative pathology show there is no lymph node metastasis (N0).

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent;
* Ability to comply with research protocols and follow-up procedures;
* The patient's age is 18 years or older;
* Histologically or cytologically confirmed as SCLC, chest-enhanced CT, liver and adrenal CT, cranial magnetic resonance, PET-CT/systemic bone imaging, etc. Definitely stage II, IIIA staged patients (according to the UICC 2009 edition staging criteria);
* Patients must have measurable lesions (according to the RECIST 1.0 standard);
* Physical status ECOG score is 0~1;
* Life expectancy is at least 12 weeks;
* The following laboratory tests were performed within 7 days prior to the first dose to confirm that the patient's bone marrow, liver, and kidney functions met the requirements for participating in the study:

  * Hemoglobin ≥ 9.0 g/dL (can be maintained or exceeded by blood transfusion);
  * The absolute neutrophil count (ANC) ≥ 1.5 × 109;
  * platelet count ≥100×109/mm3;
  * Total bilirubin ≤ 1.5 times the upper limit of normal;
  * Alanine aminotransferase and aspartate aminotransferase ≤2.5 times the normal upper limit;
  * creatinine ≤ 1.5 times the upper limit of normal; and creatinine clearance ≥ 60 ml/min;
  * The international normalized prothrombin time ratio (INR) is less than 1.5 in patients who have not received anticoagulant therapy, and the partial thromboplastin time (APTT) is less than 1.5 times the upper limit of normal. Patients receiving full-dose or parenteral anticoagulant therapy should be stable for at least 2 weeks before entry into clinical studies, and the results of the clotting test can be entered into clinical trials within the limits of local treatment.
  * Women of childbearing age must have a pregnancy test within 7 days of starting treatment and the result is negative.
  * Men and women of appropriate age must have reliable methods of contraception prior to entering the trial and during the study until 30 days after discontinuation. Reliable contraceptive methods will be determined by the principal investigator or designated person.

Exclusion Criteria:

* Conducted any systemic anti-cancer therapy for SCLC, including cytotoxic drug therapy, targeted drug therapy, and experimental therapy;
* Surgical treatment for SCLC;
* Localized radiotherapy for SCLC;
* Patients with other than SCLC cancer in the five years prior to the start of treatment in this study. Except for cervical carcinoma in situ, cured basal cell carcinoma, bladder epithelial tumor [including Ta and Tis];
* Any unstable systemic disease (including active infections, uncontrolled high blood pressure, unstable angina, angina pectoris starting in the last 3 months, congestive heart failure (≥New York Heart Association [NYHA] Grade II), myocardial infarction (6 months prior to enrollment), severe arrhythmia requiring medication, liver, kidney, or metabolic disease;
* Has or is currently suffering from interstitial lung disease;
* There are no fully controlled eye inflammations or eye infections, or any condition that may lead to the aforementioned eye diseases;
* Human immunodeficiency virus (HIV) infection is known;
* Allergies to any of the research drugs;
* Patients who have undergone major surgery or severe trauma within the first 2 months of the first dose;
* any malabsorption;
* pregnant or lactating women;
* Other investigators think it inappropriate to join the group.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2018-10 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
5-year overall survival rate | From the completion of the intervention to 5 years.
  Five-year survival rate measures survival at 5 years after treatment.

SECONDARY OUTCOMES:
recurrence rate | In 1 year after treatment.
  Patients who develop SCLC after treatment.
resection rate | At the end of Perioperative period, an average of 2 weeks.
  Patients who are eligible to receive surgery.
tumor biological makers | At the end of Perioperative period, an average of 2 weeks
  A biomarker, or biological marker, generally refers to a measurable indicator of SCLC.
overall survival rate | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 90 months
  Patients with SCLC can die directly from that disease or from an unrelated cause (for example, a car accident). When the precise cause of death is not specified called the overall survival rate.
disease-free survival rate | From date of randomization until the date of first documented progression, whichever came first, assessed up to 40 months
  The period after curative treatment [disease eliminated] when no disease can be detected.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided